CLINICAL TRIAL: NCT04505137
Title: A Phase 1, Placebo-Controlled, Double-Blind, Dose-Escalation Study To Investigate The Safety, Tolerability, And Pharmacokinetics Of A Single Intravenous Dose Of GMA301 Injection In Healthy Volunteers
Brief Title: A Study to Investigate Safe and Tolerable Dose of GMA301 Injection in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gmax Biopharm Australia Pty Ltd. (Industry)
Collaborators: Metaclinical (Unknown); Syneos Heath (Unknown)
Responsible Party: Sponsor
Organization: Gmax Biopharm LLC. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GETA_SAD_02
Record Dates: First submitted 2020-07-31; First posted 2020-08-10 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2020-11

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: Two sequential dosing cohorts, each with 6 subjects receiving GMA301 Injection and 2 subjects receiving placebo (total of 16 subjects). The doses to be administered will be 1500 mg and 2000 mg, or matching placebo, single dosing. Each cohort will include at least 2 participants of Chinese descent, if possible.
Who Masked: Participant, Investigator
Masking Description: The subjects and the clinical personnel involved in the collection, monitoring, revision, or evaluation of AEs, or personnel who could have an impact on the outcome of the study will be blinded with respect to the subject's treatment assignment (GMA301 Injection or placebo). Blinding will be maintained at least until the clinical phase of the study is completed (i.e., when reporting and evaluation of all AEs have been completed, for all cohorts).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GMA301 1500mg Or Placebo Injection (Experimental): Two sentinel subjects (1 active and 1 placebo) will be dosed first and then reaming 6 subjects will dosed within 7 days. The dose to be administered is 1500 mg single Intravenous dose of GMA301 Injection.
  Interventions: Drug: GMA301 Injection; Other: GMA301 Placebo Injection
- GMA301 2000mg Or Placebo Injection (Experimental): Two sentinel subjects (1 active and 1 placebo) will be dosed first and then reaming 6 subjects will dosed within 7 days. The dose to be administered is 2000 mg single intravenous dose of GMA301 Injection.
  Interventions: Other: GMA301 Placebo Injection; Drug: GMA301 Injection

INTERVENTIONS:
Drug: GMA301 Injection — GMA301 Injection administered as a single dose of 1500 mg
  Arms: GMA301 1500mg Or Placebo Injection
Other: GMA301 Placebo Injection — GMA301 Injection without GMA301 administered as a single intravenous dose
Drug: GMA301 Injection — GMA301 Injection administered as a single dose of 2000 mg
  Arms: GMA301 2000mg Or Placebo Injection

SUMMARY:
This study is a single-centre, randomized, double-blind, placebo-controlled, dose escalation study to assess the safety, tolerability and PK of GMA301 Injection in healthy subjects. Two sequential dosing cohorts (at ascending dose fashion), each with 6 subjects receiving GMA301 Injection and 2 subjects receiving placebo (total of 16 subjects), will be given single doses. The doses to be administered in the two cohorts will be 1500 mg and 2000 mg respectively, or matching placebo

DETAILED DESCRIPTION:
The current study is an extension of the previous study #1010218 (ACTRN12618000121268) to further explore the safety and PK profile of GMA301 injection at higher dosage. The SRC (Safety Review Committee) will be responsible for the assessment of safety, tolerability, and PK data for each dose level and to make decisions with regards to study progression. A Statistical Analysis Plan (SAP) will be written after finalizing the protocol and prior to database lock. The SAP will detail the implementation of all the planned statistical analyses in accordance with the principal features stated in the protocol. Adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoker (no use of tobacco or nicotine products within 2 months prior to screening) with BMI > 18.5 and < 30.0 kg/m2 and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females. Each cohort will include at least 2 participants of Chinese descent, if possible.
2. Healthy as defined by:

   1. The absence of clinically significant illness and surgery within 4 weeks prior to dosing.
   2. The absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Females of childbearing potential who are sexually active with a male partner must be willing to use one of the following acceptable contraceptive methods throughout the study and for 6 months after the last study drug administration:

   1. Oral, injected, or implanted hormonal methods of contraception in combination with a barrier method;
   2. Placement of an intrauterine device (IUD) or intrauterine system (IUS) in combination with a barrier method;
   3. Sterilized male partner (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate) in combination with a barrier method;
   4. True abstinence, when this is in line with the subject's preferred and usual lifestyle.
4. Male subjects must agree to avoid causing pregnancy by using a reliable method of birth control during the study and for 6 months after study drug administration and must be willing to use one of the following acceptable contraceptives:

   1. Simultaneous use of a male condom and, for the female partner, hormonal contraceptives used since at least 4 weeks or intra-uterine contraceptive device placed since at least 4 weeks;
   2. Simultaneous use of a male condom and, for the female partner, a diaphragm or cervical cap.
5. Male subjects (including men who have had a vasectomy) with a pregnant partner must agree to use a condom from the first study drug administration until at least 6 months after study drug administration.
6. Male subjects must be willing not to donate sperm during the study and for 6 months following study drug administration.
7. Capable of consent.

Exclusion Criteria:

1. Any clinically significant abnormality at physical examination, clinically significant abnormal laboratory test results or positive test for HIV, hepatitis B, or hepatitis C found during medical screening.
2. Presence or history of any clinically significant chronic condition of the neurological, respiratory, cardiovascular, gastrointestinal, urogenital, reproductive, musculoskeletal, endocrine system or cancer.
3. Clinically significant (as judged by the investigator) presence of acute illness (e.g., gastrointestinal illness, infection such as influenza, upper respiratory tract infection) upo admission to the study site.
4. Alanine aminotransferase and/or aspartate aminotransferase above the upper limit of normal.
5. Positive urine drug screen or alcohol breath test at screening.
6. Positive pregnancy test at screening.
7. Clinically significant ECG abnormalities or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 60 or over 90 mmHg,or heart rate less than 40 or over 100 bpm) at screening. Up to 2 additional measurements may be taken after an appropriate resting interval (at least 10 minutes) at Screening to confirm eligibility.
8. History of type 1 hypersensitivity or severe cutaneous adverse reaction to any medication, or to any excipient in the formulation, or history of significant atopy.
9. Hemoglobin below lower limit of normal.
10. Women who intend to become pregnant or are lactating.
11. History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit (average weekly alcohol intake that exceeds 14 units per week (males) or 7 units (females) per week, or are unwilling to stop alcohol consumption for 24 hours prior to study drug dosing until the completion of the study (1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine;1.5 oz or 45 mL of distilled spirits).
12. History of significant drug abuse within 1 year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine (PCP), crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.
13. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to dosing, administration of a biological product in the context of a clinical research study within 90 days prior to dosing, or concomitant participation in an investigational study involving no drug or device administration.
14. Use of prescription medications or over-the-counter medications within 7 days prior to study drug administration, with the exception of simple analgesics such as paracetamol and routine vitamins.
15. Donated more than 500 mL of blood within 4 weeks prior to study enrollment, or donated plasma or participated in a plasmapheresis program within 7 days of study drug administration.
16. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | All AEs (adverse events) will be captured from the time the investigator received the signed ICF (informed consent form) of subjects until study completion ie Day 70
  To assess the safety and tolerability of GMA301 Injection following single escalating intravenous (IV) injections in healthy subjects.

SECONDARY OUTCOMES:
Pharmacokinetics Profile | Blood PK samples will be collected for analysis during the treatment period at: pre-dose and 4 hours, 8 hours, 24 hours, 72 hours, 168 hours post-dose (Day 7), Day 14, Day 21, Day 28, Day 42, Day 56 and Day 70
  PK parameters determined is AUC(0-inf)
Pharmacokinetics Profile | Blood PK samples will be collected for analysis during the treatment period at: pre-dose and 4 hours, 8 hours, 24 hours, 72 hours, 168 hours post-dose (Day 7), Day 14, Day 21, Day 28, Day 42, Day 56 and Day 70
  PK parameters determined is AUC(0-t)
Pharmacokinetics Profile | Blood PK samples will be collected for analysis during the treatment period at: pre-dose and 4 hours, 8 hours, 24 hours, 72 hours, 168 hours post-dose (Day 7), Day 14, Day 21, Day 28, Day 42, Day 56 and Day 70
  PK parameters determined is C(max)
Pharmacokinetics Profile | Blood PK samples will be collected for analysis during the treatment period at: pre-dose and 4 hours, 8 hours, 24 hours, 72 hours, 168 hours post-dose (Day 7), Day 14, Day 21, Day 28, Day 42, Day 56 and Day 70
  PK parameters determined is residual area
Pharmacokinetics Profile | Blood PK samples will be collected for analysis during the treatment period at: pre-dose and 4 hours, 8 hours, 24 hours, 72 hours, 168 hours post-dose (Day 7), Day 14, Day 21, Day 28, Day 42, Day 56 and Day 70
  PK parameters determined is T(max)
Pharmacokinetics Profile | Blood PK samples will be collected for analysis during the treatment period at: pre-dose and 4 hours, 8 hours, 24 hours, 72 hours, 168 hours post-dose (Day 7), Day 14, Day 21, Day 28, Day 42, Day 56 and Day 70
  PK parameters determined is T(1/2 el)
Pharmacokinetics Profile | Blood PK samples will be collected for analysis during the treatment period at: pre-dose and 4 hours, 8 hours, 24 hours, 72 hours, 168 hours post-dose (Day 7), Day 14, Day 21, Day 28, Day 42, Day 56 and Day 70
  PK parameters determined is K(el)
Dose for GMA301 Injection for subsequent clinical studies | All AEs will be captured from the time the investigator received the signed ICF of subjects until study completion ie Day 70
  To identify appropriate doses of GMA301 Injection for subsequent clinical studies

CONTACTS AND LOCATIONS:
Overall Officials: Sepehr Shakib, Dr, Principal Investigator — CMAX Clinical Research
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No